CLINICAL TRIAL: NCT07340203
Title: Cross-Cultural Adaptation, Validity, and Reliability of the Wexner Questionnaire
Brief Title: Cross-Cultural Adaptation, Validity, and Reliability of the Wexner Questionnaire in Patients With Constipation
Status: Active, not recruiting | Type: Observational
Sponsor: Ahi Evran University Education and Research Hospital (Other)
Responsible Party: Principal Investigator, Esra BAYRAMOĞLU DEMİRDÖĞEN, Lecturer Doctor, Ahi Evran University Education and Research Hospital
Other Study IDs: KAEU-EBAYRAMOGLUD-003
Record Dates: First submitted 2025-10-28; First posted 2026-01-14 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Constipation - Functional
MeSH Terms: interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Other: survey — survey application
  Other Names: questionnaire

SUMMARY:
The investigators will conduct a validity and reliability study of the Wexner Constipation Questionnaire, used for constipation, in Turkish. For this purpose, investigators will administer the Wexner Questionnaire, translated from English to Turkish, and the accompanying Constipation Quality of Life Scale to 200 participants. Investigators will repeat the Wexner questionnaire for some participants after two weeks.

DETAILED DESCRIPTION:
To assess the cultural adaptation, validity, and reliability of the eight-question Wexner Constipation Questionnaire, the questionnaire was first translated from English to Turkish, then back from Turkish to English, and finally back from English to Turkish. The questionnaire was finalized with the collaboration of an internal medicine specialist and a gastroenterologist to prepare the Turkish version. It will then be administered to a minimum of 200 participants, along with the Constipation Quality of Life Questionnaire, previously validated and reliable in Turkish and used for constipation. For reliability, the questionnaire will be repeated for a portion of the participants after two weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Being over 18 years of age
2. Being diagnosed with functional constipation according to Rome IV criteria
3. Having undergone an anorectal examination by a gastroenterologist
4. Having no history of neurodegenerative disease (e.g., multiple sclerosis, spinal cord injury, or stroke)
5. Having no history of metabolic disorders (e.g., diabetes, hypothyroidism, or hypercalcemia)
6. Having no history of opioid-induced constipation
7. Having no history of irritable bowel syndrome
8. Having no history of congenital anorectal abnormality
9. Having no history of colon cancer or pregnancy
10. Having the ability to read and write Turkish.

Exclusion Criteria:

1. Not wanting to continue the study.
2. Having any complaints, such as anorectal bleeding, during the test-retest interval.

Ages: 18 Years to 90 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Men and women with chronic constipation
Sampling Method: Probability Sample
Enrollment: 202 (Actual)
Dates: Start 2025-07-01 (Actual); Primary Completion 2025-12-12 (Actual); Study Completion 2026-05-25 (Estimated)

PRIMARY OUTCOMES:
Application of survey to participants | approximately 1 month
  First administration of the Wexner questionnaire to all participants
Application of survey to participants | approximately 1 month
  First administration of the quality of life questionnaire to all participants

SECONDARY OUTCOMES:
Application of survey to participants | approximately 1 week
  Wexner questionnaire were administered to the participants a second time two weeks later.
Application of survey to participants | approximately 1 week
  Quality of life questionnaire were administered to the participants a second time two weeks later.

CONTACTS AND LOCATIONS:
Locations (1):
- Kirşehir Ahi Evran University Physical Therapy and Rehabilitation Hospital, Kırşehir, Centre, Turkey (Türkiye)